CLINICAL TRIAL: NCT07088913
Title: An Open-label, Fixed-sequence Study to Assess the Effect of Capivasertib on the Pharmacokinetics of Oral Rosuvastatin (a BCRP, OATP1B1 and OATP1B3 Sensitive Substrate) in Healthy Participants
Brief Title: A Study to Investigate the Effect of Capivasertib on the Pharmacokinetics of Oral Rosuvastatin in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: D3615C00006
Record Dates: First submitted 2025-07-17; First posted 2025-07-28 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Healthy Participants
Keywords: Drug-drug interaction; Pharmacokinetics; Breast Cancer Resistance Protein
MeSH Terms: interventions — capivasertib; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rosuvastatin/Capivasertib+Rosuvastatin (Experimental): Participants will receive a single dose of rosuvastatin in Period 1. After a minimum washout period of 7 days from the first dose of rosuvastatin, participants will receive the first dose of capivasertib, administered concomitantly with a single dose of rosuvastatin in Period 2, followed by a second dose of capivasertib after 12 hours.
  Interventions: Drug: Capivasertib; Drug: Rosuvastatin

INTERVENTIONS:
Drug: Capivasertib — Capivasertib will be administered orally twice in Period 2.
  Other Names: AZD5363
Drug: Rosuvastatin — Rosuvastatin will be administered orally once in both Period 1 and Period 2.
  Other Names: CRESTOR

SUMMARY:
The purpose of the study is to assess the effect of capivasertib on the pharmacokinetics (PK) of oral rosuvastatin in healthy participants.

DETAILED DESCRIPTION:
This study is an open-label, fixed-sequence, drug-drug interaction study of orally administered rosuvastatin in the presence and absence of capivasertib in healthy participants.

The study will comprise:

1. A Screening Period of maximum 28 days.
2. Two Treatment Periods

   * Period 1: Participants will receive single oral dose of rosuvastatin.
   * Period 2: Participants will receive two single oral doses of capivasertib administered 12 hours apart, with the first capivasertib dose being concomitantly administered with a single oral dose of rosuvastatin.
3. A final Follow-up Visit within 7 to 10 days after the last study intervention administration.

There will be a minimum washout period of at least 7 days between the first dose of rosuvastatin (in Treatment Period 1) and the second dose of rosuvastatin (in Treatment Period 2).

ELIGIBILITY:
Key Inclusion Criteria:

1. Healthy male and/or female participants with suitable veins for cannulation or repeated venipuncture.
2. Body Mass Index (BMI) between 18 and 32 kg/m² inclusive and weigh at least 50 kg and no more than 150 kg inclusive.
3. All females must have a negative pregnancy test at the Screening Visit and on admission to the Clinical Unit and must not be lactating.
4. Females of non-childbearing potential must be confirmed at the Screening Visit by fulfilling one of the following criteria:

   1. Postmenopausal (≥12 months of amenorrhea + hormone confirmation).
   2. Irreversible surgical sterilization by hysterectomy and/or bilateral oophorectomy, and/or bilateral salpingectomy (excluding tubal ligation) at least 6 months prior to screening.
5. Male participants must be vasectomized (at least 6 months prior to screening), with documented post-procedural medical assessment of surgical success.
6. Participants must be willing to use study-specific contraceptive methods.

Key Exclusion Criteria:

1. History of any clinically important disease or disorder which may either put the participant at risk because of participation in the study or influence the results or the participant's ability to participate in the study.
2. History or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
3. Any clinically important illness, medical/surgical procedure, or trauma.
4. Any clinically significant skin abnormalities that are chronic or currently active.
5. Any clinically important abnormalities in clinical chemistry, hematology, or urinalysis results.
6. Any positive result on screening for serum Hepatitis B surface antigen (HBsAg), Hepatitis B core antibody (HBcAb), Hepatitis C virus antibody (HCV antibody), or Human Immunodeficiency Virus (HIV).
7. Any clinically significant abnormalities in blood lipid profiles (triglycerides, high-density lipoprotein, low-density lipoprotein, and total cholesterol).
8. Any clinically significant abnormalities in glucose metabolism, including:

   1. Diagnosis of type I or II diabetes mellitus (irrespective of management),
   2. Fasting blood glucose ≥ 100 mg/dL, or
   3. Hemoglobin A1c > 5.7% after at least 8 hours of fasting at screening.
9. Any clinically significant abnormal findings in vital signs.
10. Any clinically significant abnormalities on 12-lead electrocardiogram (ECG) and defined as Sick sinus syndrome, arrhythmia, prolonged QTcF > 450 ms, family history of long QT syndrome, persistent or intermittent bundle branch block, and atrio-ventricular block Grade II or III.
11. Current smokers or those who have smoked or used nicotine products (including e-cigarettes) within the previous 3 months.
12. Known or suspected history of alcohol or drug abuse or excessive intake of alcohol.
13. History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity or history of hypersensitivity to drugs with a similar chemical structure or class to capivasertib or rosuvastatin or history of hypersensitivity to any component of the finished dosage form of capivasertib.
14. Plasma donation or any blood donation/blood loss prior to the Screening Visit.
15. Participants who have previously received capivasertib.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2026-03-26 (Estimated); Study Completion 2026-03-26 (Estimated)

PRIMARY OUTCOMES:
Area under concentration-time curve from time 0 to infinity (AUCinf) of rosuvastatin | Period 1: Day 1 to Day 3 and Period 2: Day 1 to Day 3
  To evaluate the PK (AUCinf) of rosuvastatin when administered orally alone and in combination with capivasertib.
Area under concentration-curve from time 0 to the last quantifiable concentration (AUClast) of rosuvastatin | Period 1: Day 1 to Day 3 and Period 2: Day 1 to Day 3
  To evaluate the PK (AUClast) of rosuvastatin when administered orally alone and in combination with capivasertib.
Maximum observed drug concentration (Cmax) of rosuvastatin | Period 1: Day 1 to Day 3 and Period 2: Day 1 to Day 3
  To evaluate the PK (Cmax) of rosuvastatin when administered orally alone and in combination with capivasertib.

SECONDARY OUTCOMES:
Ratio of AUCinf (R AUCinf) of rosuvastatin | Period 1: Day 1 to Day 3 and Period 2: Day 1 to Day 3
  To evaluate the PK (R AUCinf) of rosuvastatin when administered orally alone and in combination with capivasertib.
Ratio of AUClast (R AUClast) of rosuvastatin | Period 1: Day 1 to Day 3 and Period 2: Day 1 to Day 3
  To evaluate the PK (R AUClast) of rosuvastatin when administered orally alone and in combination with capivasertib.
Ratio of Cmax (R Cmax) of rosuvastatin | Period 1: Day 1 to Day 3 and Period 2: Day 1 to Day 3
  To evaluate the PK (R Cmax) of rosuvastatin when administered orally alone and in combination with capivasertib.
Terminal elimination half-life (t½λz) of rosuvastatin | Period 1: Day 1 to Day 3 and Period 2: Day 1 to Day 3
  To evaluate the PK (t½λz) of rosuvastatin when administered orally alone and in combination with capivasertib.
Terminal elimination rate constant (λz) of rosuvastatin | Period 1: Day 1 to Day 3 and Period 2: Day 1 to Day 3
  To evaluate the PK (λz) of rosuvastatin when administered orally alone and in combination with capivasertib.
Time to reach maximum observed concentration (tmax) of rosuvastatin | Period 1: Day 1 to Day 3 and Period 2: Day 1 to Day 3
  To evaluate the PK (tmax) of rosuvastatin when administered orally alone and in combination with capivasertib.
AUClast of capivasertib | Period 2: Day 1 to Day 3
  To evaluate the PK (AUClast) of capivasertib following oral dosing.
Concentration at the end of a dosing interval (Ctrough) of capivasertib | Period 2: Day 1 to Day 3
  To evaluate the PK (Ctrough) of capivasertib following oral dosing.
Cmax of capivasertib | Period 2: Day 1 to Day 3
  To evaluate the PK (Cmax) of capivasertib following oral dosing.
Number of participants with adverse events (AEs) and serious AEs | From Screening (Day -30 to Day -2) to follow-up visit (Day 10)
  To assess the safety and tolerability of capivasertib when administered with rosuvastatin.
Change in serum bilirubin levels | Day 1 (pre-capivasertib dose) to Day 3 (post-capivasertib dose)
  To evaluate the effect of capivasertib dosing on total, conjugated, and unconjugated bilirubin levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/